CLINICAL TRIAL: NCT03712137
Title: A Multicenter, Evaluator-blinded, Randomized, Parallel-group, Controlled Study of the Safety and Effectiveness of JUVÉDERM VOLUX™ XC Injectable Gel for Restoring Jawline Definition
Brief Title: Study of the Safety and Effectiveness of JUVÉDERM VOLUX™ XC Injectable Gel for Restoring Jawline Definition
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: V25L-002
Record Dates: First submitted 2018-10-17; First posted 2018-10-19 (Actual); Results first posted 2023-01-04 (Actual); Last update posted 2023-01-04 (Actual); Status verified 2022-09

CONDITIONS: Jawline Definition

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- VOLUX XC (Experimental): Participants will be treated with VOLUX XC hyaluronic acid (HA) injectable gel on day 1 with optional touch-up at day 30 and optional maintenance treatment at Month 12.
  Interventions: Device: VOLUX XC
- No-treatment control (Experimental): No-treatment during the control period. Optional delayed-treatment with VOLUX XC (initial with optional touch-up) at the beginning of the Post-Control period.
  Interventions: Other: No-treatment control

INTERVENTIONS:
Device: VOLUX XC — Participants will be treated with VOLUX XC hyaluronic acid (HA) injectable gel on day 1 with optional touch-up at day 30 and optional maintenance treatment at Month 12.
  Arms: VOLUX XC
Other: No-treatment control — No-treatment during the control period. Optional delayed-treatment with VOLUX XC (initial with optional touch-up) at the beginning of the Post-Control period.
  Arms: No-treatment control

SUMMARY:
This study will evaluate the safety and effectiveness of JUVÉDERM VOLUX™ XC injectable gel for restoring jawline definition

ELIGIBILITY:
Inclusion Criteria:

* Has "Moderate" or "Severe" loss of jawline definition as determined by the EI using the ALJDs (Grade 2 or 3 on the ALJDS) on both sides. The grade does not have to be the same on both sides, but must be Grade 2 or 3
* Treating Investigator (TI) considers the subject's jaw amenable to an improvement of at least 1 grade on the scale for the jawline definition
* Written Informed Consent (IC) has been obtained

Exclusion Criteria:

* Has ever received permanent facial implants (eg, polymethylmethacrylate, silicone, polytetrafluoroethylene) anywhere in the face or neck, or is planning to be implanted with any of these products during the study
* Has ever undergone fat injections in the malar, chin or jawline area or is planning to undergo this procedure during the study
* Has undergone semipermanent dermal filler treatment (eg, calcium hydroxyapatite, poly-L-lactic acid) below the subnasale within 36 months before enrollment or is planning to undergo such treatment during the study
* Has received deoxycholic acid treatment in the submental region in the last 6 months
* Has active autoimmune disease
* Females who are pregnant, nursing, or planning a pregnancy during the course of the study

Min Age: 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 206 (Actual)
Dates: Start 2018-11-12 (Actual); Primary Completion 2020-02-04 (Actual); Study Completion 2021-01-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marta Sartor, Study Director — Allergan
Locations (19):
- United States (19):
  - Total Skin and Beauty Dermatology Center, PC, Birmingham, Alabama
  - Westside Aesthetics, Los Angeles, California
  - Artemedica, Santa Rosa, California
  - Center for Dermatology and Dermatologic Surgery, Washington D.C., District of Columbia
  - Susan H Weinkle, MD, Bradenton, Florida
  - Hevia Cosmetic Dermatology, Coral Gables, Florida
  - Skin Research Institute LLC, Coral Gables, Florida
  - Baumann Cosmetic and Research Institute, Miami, Florida
  - DeNova Research dba Arano, LLC, Chicago, Illinois
  - Callender Center for Clinical Research, Glenn Dale, Maryland
  - MDLSV, Hunt Valley, Maryland
  - Williams Center, Latham, New York
  - The Center for Dermatology, Cosmetic & Laser Surgery, Mount Kisco, New York
  - Center aesthetic and dermatology, New York, New York
  - Laser & Skin Surgery Center of New York, New York, New York
  - Aesthetic Solutions, PA., Chapel Hill, North Carolina
  - Bellaire Dermatology Associates, Bellaire, Texas
  - Suzanne Bruce and Associates, P.A., The Center for Skin Research, Houston, Texas
  - SkinDC, Arlington, Virginia

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study consists of 2 groups: Treatment and Control. The treatment group rec'd treatment Day 1 and was followed up to Month 12. At Month 12 they had the option to exit the study or receive maintenance treatment with an add'l 3 months of follow-up after treatment. The control group followed a 6-month no-treatment control period after which they had the option to exit the study or proceed to the post-control period where they receive treatment with 12 months of follow-up after their last treatment.
Groups:
- No-treatment Control: No-treatment at the beginning of the control period. Optional delayed-treatment with VOLUX XC (initial with optional touch-up) during the Post-Control period.
  No-treatment control: No-treatment during the control period. Optional delayed-treatment with VOLUX XC (initial with optional touch-up) during the Post-Control period.
Period: Control Period
Arm/Group | No-treatment Control | VOLUX XC
Started | 49 | 157
Participants Treated as Randomized | 49 | 156
Participants Not Treated as Randomized (Participant was randomized to the treatment group (VOLUX XC) but subsequently found to not meet inclusion criteria and was discontinued at randomization without receiving treatment.) | 0 | 1
Completed | 47 | 149
Not Completed | 2 | 8
Period: Opt VOLUX Treatment Follow Up Period
Arm/Group | No-treatment Control | VOLUX XC
Started (Participants that were randomized to the No-Treatment Control arm that received optional VOLUX treatment after the Control Period) | 42 | 0
Completed | 35 | 0
Not Completed | 7 | 0
Period: VOLUX Maintenance Treatment Period
Arm/Group | No-treatment Control | VOLUX XC
Started (Participants in the VOLUX XC treatment population who received VOLUX maintenance treatment) | 0 | 87
Completed | 0 | 85
Not Completed | 0 | 2

BASELINE CHARACTERISTICS:
Population: Modified intent-to-treat (mITT) Population included all randomized participants with non-missing baseline on the ALJDS scale on both sides of the jaw
Groups:
- Total: Total of all reporting groups
Arm/Group | No-treatment Control | VOLUX XC | Total
Number analyzed (Participants) | 49 | 157 | 206
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.9 (9.37) | 59.3 (8.22) | 59.0 (8.50)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39 | 141 | 180
  Male | 10 | 16 | 26
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 11 | 31 | 42
  Not Hispanic or Latino | 38 | 126 | 164
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 21 | 27
  White | 42 | 132 | 174
  More than one race | 1 | 3 | 4
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 49 | 157 | 206
Participant Level Allergan Loss of Jawline Definition Scale (ALJDS) [Number; unit: units on a scale] — If the baseline ALJDS score is different for left and right jaws, then the participant is included under the worse score.
  units on a scale
    Moderate | 13 | 34 | 47
    Severe | 36 | 114 | 150
    Extreme | 0 | 9 | 9

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Show ≥ 1-point Jawline Improvement on Both Sides From Baseline on the Allergan Loss of Jawline Definition Scale (ALJDS)
Description: The ALJDS is an Investigator assessment of loss of jawline definition measured by a 5-point scale (0=None, 1=Mild, 2=Moderate, 3=Severe, 4=Extreme)
Time Frame: Month 6
Population: All modified intent-to-treat (mITT) participants who have Month 6 assessment on the ALJDS scale on both sides of the jaw. Multiple imputation was performed on participants with missing data for the Month 6 assessment on the ALJDS on both sides of jaw
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | No-treatment Control | VOLUX XC
Number analyzed (Participants) | 49 | 157
percentage of participants | 38.0 [24.25 to 51.80] | 69.0 [61.53 to 76.39]
Statistical Analysis 1: Comparison: VOLUX XC; Test type: Superiority; p = 0.0001, Multiple Imputation; The procedure used to perform Multiple Imputation is PROC MIANALYZE in SAS with normal approximation; Responder Rate Difference = 30.9, 95% CI 2-sided [15.33 to 46.54]

2. Secondary Outcome: Percentage of Participants Who Note "Improved" or "Much Improved" in Jawline Area as Assessed by the Evaluating Investigator Using the Global Aesthetic Improvement Scale (GAIS)
Description: The Evaluating Investigator (EI) will assess the aesthetic improvement of the jawline area using the GAIS 5-point scale where: 2=much improved, 1=improved, 0=no change, -1=worse and -2=much worse. The percentage of participants who the Evaluating Investigator assesses as 2=much improved or 1=improved will be reported.
Time Frame: Month 6
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | No-treatment Control | VOLUX XC
Number analyzed (Participants) | 45 | 146
Participants | 13 | 130

3. Secondary Outcome: Percentage of Participants Who Note "Improved" or "Much Improved" in Jawline Area as Assessed by the Participant Using the Global Aesthetic Improvement Scale (GAIS)
Description: The participant will assess the aesthetic improvement of the jawline area using the GAIS 5-point scale where: 2=much improved, 1=improved, 0=no change, -1=worse and -2=much worse. The percentage of participants who assess themselves as 2=much improved or 1=improved will be reported.
Time Frame: Month 6
Population: As per the Protocol and the Statistical Analysis Plan: During the Control Period these data were collected only for participants that were randomized and received VOLUX treatment at the beginning of the Control Period
Measure: Count of Participants; unit: Participants
Arm/Group | VOLUX XC
Number analyzed (Participants) | 146
Participants | 129

4. Secondary Outcome: Change From Baseline in Overall Score for FACE-Q™ Satisfaction With Lower Face and Jawline Score
Description: The subject will assess satisfaction using the 5 questions on the Satisfaction of Lower Face and Jawline scale of the FACE-Q™ questionnaire measured on a 4-point scale (1=Very Dissatisfied 2=Somewhat Dissatisfied, 3=Somewhat Satisfied, 4=Very Satisfied). The raw scale summed score will then be converted into a Rasch-transformed score from 0 (worst) to 100 (best)
Time Frame: Baseline to Month 6
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | VOLUX XC
Number analyzed (Participants) | 146
score on a scale | 45.9 (33.09)
Statistical Analysis 1: Comparison: VOLUX XC; Test type: Superiority; p < 0.0001, Paired T-test; Mean Difference (Final Values) = 45.9, 95% CI 2-sided [40.45 to 51.28]

ADVERSE EVENTS:
Time Frame: 12 to 17 months for the treatment group and 6 to 20 months for the control group.
Description: All randomized participants who receive study treatment (VOLUX or control) make up the Safety Population. There is one participant, that was randomized in error, that did not receive the treatment and is assigned to the control treatment arm for reporting purposes.
Groups:
- No-treatment Control: No-treatment during the control period.
  No-treatment control: No-treatment during the control period. (randomization to Month 6)
- VOLUX XC Treatment: Participants will be treated with VOLUX XC hyaluronic acid (HA) injectable gel on day 1 with optional touch-up at day 30 and optional maintenance treatment at Month 12.
  VOLUX XC: Participants will be treated with VOLUX XC hyaluronic acid (HA) injectable gel on day 1 with optional touch-up at day 30 and optional maintenance treatment at Month 12.
- Optional VOLUX XC Treatment Post Control: Optional delayed-treatment with VOLUX XC (initial with optional touch-up) during the Post-Control period (optional treatment to study exit).
- VOLUX Maintenance Treatment: Participants in the VOLUX XC Treatment population who received VOLUX maintenance treatment at Month 12
Arm/Group | No-treatment Control | VOLUX XC Treatment | Optional VOLUX XC Treatment Post Control | VOLUX Maintenance Treatment
All-Cause Mortality (participants affected / at risk) | 0/50 | 0/156 | 0/42 | 0/87
Serious Adverse Events (participants affected / at risk) | 1/50 | 17/156 | 3/42 | 4/87
Other Adverse Events (participants affected / at risk) | 0/50 | 9/156 | 5/42 | 1/87
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | No-treatment Control (N=50) | VOLUX XC Treatment (N=156) | Optional VOLUX XC Treatment Post Control (N=42) | VOLUX Maintenance Treatment (N=87)
INJECTION SITE HYPERSENSITIVITY (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
INJECTION SITE NODULE (General disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
BACTERIAL VAGINOSIS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
BRONCHITIS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
CELLULITIS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
CLOSTRIDIUM DIFFICILE INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
DIVERTICULITIS (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
IMPLANT SITE INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
INJECTION SITE INFECTION (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTITIS MEDIA (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
PHARYNGITIS STREPTOCOCCAL (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
SINUSITIS (Infections and infestations) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
TOOTH INFECTION (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
URINARY TRACT INFECTION (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
FOOT FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
ARTHRITIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
SPINAL OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
SCHWANNOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
TRIPLE NEGATIVE BREAST CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
BREAST NECROSIS (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | No-treatment Control (N=50) | VOLUX XC Treatment (N=156) | Optional VOLUX XC Treatment Post Control (N=42) | VOLUX Maintenance Treatment (N=87)
SEASONAL ALLERGY (Immune system disorders) | 0 (0) | 2 (2) | 3 (3) | 0 (0)
HEADACHE (Nervous system disorders) | 0 (0) | 7 (7) | 3 (3) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.

DOCUMENTS (2):
  • Study Protocol (2019-03-11): https://cdn.clinicaltrials.gov/large-docs/37/NCT03712137/Prot_000.pdf
  • Statistical Analysis Plan (2020-04-28): https://cdn.clinicaltrials.gov/large-docs/37/NCT03712137/SAP_001.pdf